CLINICAL TRIAL: NCT01512758
Title: A Phase 1 Dose Escalation and Pharmacokinetic Study of Alisertib (MLN8237), an Aurora A Kinase Inhibitor, in Adult East Asian Patients With Advanced Solid Tumors or Lymphomas
Brief Title: A Study of Alisertib (MLN8237) in Adult East Asian Participants With Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C14013; 1015004128 (Registry Identifier: TCTIN); U1111-1187-6744 (Registry Identifier: WHO)
Record Dates: First submitted 2012-01-13; First posted 2012-01-19 (Estimated); Results first posted 2019-03-15 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-11

CONDITIONS: Advanced Solid Tumors; Lymphomas
Keywords: East Asian Patients; Advanced solid tumors; Lymphomas; MLN8237; Alisertib; Aurora A Kinase Inhibitor; Drug therapy
MeSH Terms: conditions — Lymphoma | interventions — MLN 8237

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alisertib 30 mg (Experimental): Alisertib 30 mg enteric-coated tablets (ECT), orally, twice a day (BID) for 7 days, followed by a 14-day rest period, in 21-day cycles until there is evidence of disease progression or unacceptable alisertib-related toxicities (up to 16 cycles). Cycles could be extended to 28-day cycles (with additional 7-day rest period) if all alisertib-related toxicities (except alopecia) were not resolved to less than Grade 2.
  Interventions: Drug: Alisertib
- Alisertib 40 mg (Experimental): Alisertib 40 mg ECT, orally, BID for 7 days, followed by a 14-day rest period, in 21-day cycles until there is evidence of disease progression or unacceptable alisertib-related toxicities (up to 7 cycles). Cycles could be extended to 28-day cycles (with additional 7-day rest period) if all alisertib-related toxicities (except alopecia) were not resolved to less than Grade 2.
  Interventions: Drug: Alisertib

INTERVENTIONS:
Drug: Alisertib — Alisertib enteric-coated tablets
  Other Names: MLN8237

SUMMARY:
The purpose of this study was to determine the safety profile, maximum tolerated dose (MTD), recommended Phase 2 dose (RP2D), and to characterize the pharmacokinetic (PK) profile of alisertib twice daily (BID) dosing for 7 days in East Asian participants with advanced solid tumors or lymphomas. The secondary objective was to describe any antitumor activity that may have been observed with alisertib treatment.

DETAILED DESCRIPTION:
The drug being tested in this study is called alisertib (MLN8237). Alisertib is being tested to treat people who have advanced solid tumors or lymphomas for which standard curative or life-prolonging treatment did not exist or was no longer effective or tolerable. This study evaluated the safety and pharmacokinetic (PK) profile, and maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of alisertib, as well as any antitumor activity.

The study enrolled 36 patients. Participants were assigned to one of the two treatment groups and received:

* Alisertib 30 mg
* Alisertib 40 mg All participants took two enteric-coated tablets every 12 hours each day for 7 days followed by a 14-day rest period in a 21-day cycle for up to 16 cycles.

This multi-center trial is conducted in East Asia. The overall time to participate in this study was 24 months, unless it was determined that a participant would derive benefit from continued therapy beyond 24 months. Participants made multiple visits to the clinic, and were contacted up to a maximum of 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female East Asian participants 18 years or older
* Histologically or cytologically confirmed metastatic and/or advanced solid tumors or lymphomas for which no effective standard treatment is available
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Expected survival longer than 3 months from study enrollment
* Radiographically or clinically evaluable tumor
* Female participants who are post menopausal for at least 1 year, surgically sterile, or agree to practice 2 effective methods of contraception through 30 days after the last dose of study drug or agree to abstain from heterosexual intercourse
* Male participants who agree to practice effective barrier contraception through 6 months after the last dose of alisertib or agree to abstain from heterosexual intercourse
* Voluntary written consent

Exclusion Criteria:

* Female participants who are lactating or pregnant
* Treatment with any investigational products, systemic antineoplastic treatment, or antineoplastic treatment with glucocorticoids within 21 days preceding the first dose of alisertib
* Treatment with nitrosoureas, mitomycin C, rituximab, alemtuzumab, or other unconjugated antibody treatment within 42 days (21 days if clear evidence of progressive disease)
* Medical conditions requiring daily, chronic, or regular use of proton pump inhibitors or H2-receptor antagonists
* Treatment with radioimmunoconjugates such as ibritumomab tiuxetan or tositumomab within 56 days preceding first alisertib dose
* Major surgery within the 14 days preceding the first dose of alisertib
* Life-threatening or uncontrolled medical illness unrelated to cancer
* Known gastrointestinal (GI) disease or procedures that could interfere with the oral absorption or tolerance of alisertib
* Inability to swallow capsules
* Inadequate bone marrow or other organ function
* Diagnosed or treated for another malignancy within 2 years of first dose of alisertib, or previously diagnosed with another malignancy and have any radiographic or biochemical marker evidence of active disease. In the case of prior prostate cancer treated with radiotherapy, the prostate specific antigen (PSA) may be detectable, but must be < 1 ng/mL. Participants with completely resected basal cell carcinoma, squamous cell carcinoma of the skin, or in situ malignancy of any type are not excluded
* Other severe acute or chronic medical or psychiatric conditions, including uncontrolled diabetes, or laboratory abnormality
* Known or suspected human immunodeficiency virus (HIV) positive or hepatitis B surface antigen-positive status, or known or suspected active hepatitis C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02-06 (Actual); Primary Completion 2013-10-08 (Actual); Study Completion 2013-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- National Cancer Centre, Tiong Bahru, Singapore

REFERENCES:
- [Derived] Venkatakrishnan K, Kim TM, Lin CC, Thye LS, Chng WJ, Ma B, Chen MH, Zhou X, Liu H, Kelly V, Kim WS. Phase 1 study of the investigational Aurora A kinase inhibitor alisertib (MLN8237) in East Asian cancer patients: pharmacokinetics and recommended phase 2 dose. Invest New Drugs. 2015 Aug;33(4):942-53. doi: 10.1007/s10637-015-0258-y. Epub 2015 Jun 19. PMID 26084989

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 8 investigative sites in Singapore, Taiwan, Hong Kong, and South Korea from 06 February 2012 to 08 October 2013.
Pre-assignment Details: Participants with a diagnosis of advanced solid tumors or lymphomas received alisertib 30 mg or 40 mg twice a day (BID) for 7 consecutive days followed by a 14-day rest period in 21-day cycles (28-day cycles with additional 7-day rest period if all alisertib-related toxicities [except alopecia] were not resolved to less than Grade 2).
Period: Overall Study
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Started | 30 | 6
Completed | 30 (Completed=Completed protocol-specified dosing and PK assessment.) | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population is defined as all participants who received at least one dose of alisertib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alisertib 30 mg | Alisertib 40 mg | Total
Number analyzed (Participants) | 30 | 6 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (9.52) | 50.7 (18.25) | 56.1 (11.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 13
  Male | 19 | 4 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian (Chinese) | 17 | 5 | 22
  Asian (Korean) | 13 | 0 | 13
  Malay | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 30 | 6 | 36
Region of Enrollment [Count of Participants; unit: Participants]
  Singapore | 4 | 6 | 10
  Taiwan | 8 | 0 | 8
  Hong Kong | 5 | 0 | 5
  Korea, Republic of | 13 | 0 | 13
Height [Mean (Standard Deviation); unit: cm] | 162.5 (6.84) | 161.9 (6.61) | 162.4 (6.71)
Weight [Mean (Standard Deviation); unit: kg] | 57.78 (9.255) | 62.30 (11.714) | 58.53 (9.669)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m^2] — BSA = square root [height (cm) x weight (kg)/3600]
  m^2 | 1.611 (0.1487) | 1.667 (0.1613) | 1.620 (0.1499)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D)
Description: MTD was defined as highest dose at which <2 participants experienced a dose-limiting toxicity (DLT). DLT was defined as any of the following events considered possibly related to therapy with alisertib by the investigator: 1. Grade 4 neutropenia (absolute neutrophil count <500 cells/mm^3) for >7 days; 2. Grade 4 neutropenia with fever (oral or ear temperature ≥38.5°C); 3. Grade 4 thrombocytopenia (platelets <25,000/mm^3) for >7 days; 4. Platelet count <10,000 cells/mm^3; 5. ≥Grade 3 thrombocytopenia with clinically significant bleeding; 6. Delay in initiation of subsequent cycle by >7 days due to treatment-related toxicity; 7. ≥Grade 3 nonhematological toxicity except following: a. ≥Grade 3 nausea and/or emesis in the absence of optimal antiemetic therapy; b. ≥Grade 3 diarrhea in the absence of optimal supportive therapy; c. Grade 3 fatigue lasting <1 week; d. Other Grade 3 nonhematological toxicity that can be safely and reliably controlled to ≤Grade 2 with appropriate treatment.
Time Frame: Treatment Cycle 1
Population: DLT-Evaluable population is defined as participants with a common race who had not used granulocyte colony-stimulating factor (G-CSF) in cycle 1, and either experienced DLT during Cycle 1 or received at least 85% of planned doses of alisertib and have sufficient follow up data to allow investigator and sponsor to determine whether a DLT occurred.
Measure: Number; unit: mg
Groups:
- Alisertib 30 mg or 40 mg: Alisertib 30 mg or 40 mg enteric-coated tablets, orally, twice a day (BID) on Days 1 through 7, followed by a 14-day rest period, in a 21-day cycle (28-day cycle with additional 7-day rest period if all alisertib-related toxicities [except alopecia] were not resolved to less than Grade 2), for a maximum of 24 months or until there is evidence of disease progression or unacceptable treatment related toxicity (up to 16 cycles).
Arm/Group | Alisertib 30 mg or 40 mg
Number analyzed (Participants) | 8
mg | 30

2. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A Serious Adverse Event (SAE) A serious is any experience that suggests a significant hazard, contraindication, side effect or precaution that: results in death, is life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or is medically significant.
Time Frame: First dose to 30 days past last dose (Up to 12.1 Months)
Population: Safety Population is defined as all participants who received at least one dose of alisertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 30 | 6
Participants
  AE | 30 | 6
  SAE | 15 | 4

3. Primary Outcome: Number of Participants With Abnormal Clinical Laboratory Values Reported as Adverse Events
Description: Laboratory AEs in the following system organ classes (SOCs) are reported: blood and lymphatic system disorders, investigations, and metabolism and nutrition disorders. An abnormal laboratory value was assessed as an AE if that value lead to discontinuation or delay in treatment, dose modification, therapeutic intervention, or was considered by the investigator to be a clinically significant change from baseline. A treatment¬-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: First dose to 30 days past last dose (Up to 12.1 Months)
Population: Safety Population is defined as all participants who received at least one dose of alisertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 30 | 6
Participants
  Neutropenia | 19 | 5
  Anaemia | 9 | 4
  Thrombocytopenia | 6 | 1
  Febrile neutropenia | 4 | 1
  Leukopenia | 2 | 2
  White blood cell count decreased | 7 | 0
  Aspartate aminotransferase increased | 6 | 0
  Neutrophil count decreased | 4 | 0
  Alanine aminotransferase increased | 4 | 0
  Platelet count decreased | 3 | 0
  Blood bilirubin increased | 2 | 0
  Haemoglobin decreased | 1 | 0
  Blood creatinine increased | 0 | 1
  Urine output decreased | 1 | 0
  Hypokalaemia | 4 | 3
  Hypercalcaemia | 0 | 1
  Hyponatraemia | 1 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs Reported as Adverse Events
Description: Vital signs (blood pressure, pulse rate, and oral temperature) measurements were collected throughout the study.
Time Frame: First dose to 30 days past last dose (Up to 12.1 Months)
Population: Safety Population is defined as all participants who received at least one dose of alisertib.
Measure: Count of Participants; unit: Participants
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 30 | 6
Participants
  Hypertension | 1 | 0
  Hypotension | 1 | 0
  Bradycardia | 1 | 0
  Pyrexia | 8 | 1

5. Primary Outcome: Cmax: Maximum Observed Concentration for Alisertib
Time Frame: Cycle 1 Days 1 and 7 predose and at multiple time points (up to 12 hours) postdose
Population: Pharmacokinetic (PK) Population is defined as all participants with sufficient dosing and PK concentration time data to reliably estimate PK parameters. "n" in the category is the number of participants with data available at the given time-point.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 30 | 6
nM
  Day 1 | 1442.5 (534.80) | 1871.7 (429.62)
  Day 7: number analyzed (Participants) | 28 | 6
  Day 7 | 3000.0 (1329.38) | 3686.7 (885.45)

6. Primary Outcome: Tmax: Time to First Occurrence of Cmax for Alisertib
Time Frame: Cycle 1 Days 1 and 7 predose and at multiple time points (up to 12 hours) postdose
Population: PK Population is defined as all participants with sufficient dosing and PK concentration time data to reliably estimate PK parameters. "n" in the category is the number of participants with data available at the given time-point.
Measure: Median (Full Range); unit: hr
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 30 | 6
hr
  Day 1 | 3.0 [2 to 8] | 2.0 [2 to 3]
  Day 7: number analyzed (Participants) | 28 | 6
  Day 7 | 2.9 [1 to 6] | 2.0 [1 to 3]

7. Primary Outcome: AUCτ: Area Under the Concentration-Time Curve From Time 0 to End of Dosing Interval (τ) for Alisertib
Time Frame: Cycle 1 Days 1 and 7 predose and at multiple time points (up to 12 hours) postdose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nM*hr
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 30 | 6
nM*hr
  Day 1 | 9549.0 (4119.30) | 11811.7 (2845.76)
  Day 7: number analyzed (Participants) | 28 | 6
  Day 7 | 24377.9 (13261.61) | 30683.3 (9575.68)

8. Primary Outcome: Dose Normalized AUCτ: Area Under the Concentration-Time Curve From Time 0 to Time t for Alisertib
Description: Dose normalized AUCτ was obtained using AUCτ divided by alisertib dose in milligrams.
Time Frame: Cycle 1 Day 7 predose and at multiple time points (up to 12 hours) postdose
Population: PK Population is defined as all participants with sufficient dosing and PK concentration time data to reliably estimate PK parameters.
Measure: Mean (Standard Deviation); unit: nM*hr/mg
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 28 | 6
nM*hr/mg | 812.9 (441.90) | 766.8 (238.88)

9. Primary Outcome: T1/2: Terminal Half-Life for Alisertib
Time Frame: Cycle 1 Day 7 predose and at multiple time points (up to 12 hours) postdose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 24 | 6
hr | 16.750 (8.1710) | 14.795 (4.5715)

10. Primary Outcome: Rac: Accumulation Ratio for Alisertib
Time Frame: Cycle 1 Day 7 predose and at multiple time points (up to 12 hours) postdose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 28 | 6
ratio | 2.830 (1.2955) | 2.690 (1.0638)

11. Primary Outcome: PTR: Peak Trough Ratio During a Dosing Interval, at Steady State for Alisertib
Time Frame: Cycle 1 Day 7 predose and at multiple time points (up to 12 hours) postdose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 28 | 6
ratio | 2.254 (0.6458) | 2.207 (0.3946)

12. Primary Outcome: CLss/F: Apparent Clearance After Extravascular Administration, at Steady State, Calculated Using AUCτ for Alisertib
Time Frame: Cycle 1 Day 7 predose and at multiple time points (up to 12 hours) postdose
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 28 | 6
L/hr | 2.9357 (1.37091) | 2.8083 (1.20259)

13. Secondary Outcome: Best Overall Response Rate Based on Investigator Assessment
Description: Best overall response rate is defined as the percentage of participants with complete response (CR) and/or partial response (PR) as assessed by the Investigator using Lymphoma International Working Group (IWG) Criteria or Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1 for target lesions and assessed by CT, PET or MRI. IWG criteria for CR is defined as the disappearance of all evidence of disease and PR is defined as regression of measurable disease and no new sites. RECIST response criteria is defined as: CR is defined as disappearance of all target lesions and PR is defined as 30% decrease in the sum of the longest diameter of target lesions.
Time Frame: Baseline and every 2 cycles for up to 24 months or until progressive disease
Population: Safety Population is defined as all participants who received at least one dose of alisertib.
Measure: Number; unit: percentage of participants
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 30 | 6
percentage of participants
  CR | 0 | 0
  PR | 3 | 0

14. Secondary Outcome: Duration of Response
Description: DOR is defined as the time from the date of first documentation of a CR response to the date of first documentation of PD according to IWG criteria or RECIST criteria 1.1. IWG PD is defined as PD is defined as any new lesion or increase by >50% of previously involved sites from nadir. RECIST PD is defined as unequivocal progression of existing non-target lesions.
Time Frame: First documented response until disease progression; approximately 12 months
Population: Safety Population is defined as all participants who received at least one dose of alisertib. Participants with response were evaluated.
Measure: Median (Full Range); unit: days
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 1 | 0
days | 169 [169 to 169] |

15. Secondary Outcome: Concentrations of Relevant Tumor Markers
Time Frame: Cycle 1, Day 1; at end of Cycle 2 and every 2 cycles thereafter; and at end treatment; approximately 12 months
Population: Data was not analyzed as per the change in planned analysis (protocol amendment).
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: First dose to 30 days past last dose (Up to 12.1 Months)
Description: At each visit the Investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alisertib 30 mg | Alisertib 40 mg
Serious Adverse Events (participants affected / at risk) | 15/30 | 4/6
Other Adverse Events (participants affected / at risk) | 30/30 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 30 mg (N=30) | Alisertib 40 mg (N=6)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Lower extremity mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Axillary mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — One treatment-emergent death occurred during treatment with alisertib 30 mg and was not related.
Pyrexia (General disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 3
Haematochezia (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alisertib 30 mg (N=30) | Alisertib 40 mg (N=6)
Diarrhoea (Gastrointestinal disorders) | 17 | 3
Stomatitis (Gastrointestinal disorders) | 16 | 2
Abdominal pain (Gastrointestinal disorders) | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 7 | 0
Nausea (Gastrointestinal disorders) | 6 | 1
Vomiting (Gastrointestinal disorders) | 5 | 1
Oral pain (Gastrointestinal disorders) | 2 | 2
Constipation (Gastrointestinal disorders) | 3 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 2
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 0
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 19 | 3
Anaemia (Blood and lymphatic system disorders) | 8 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1
Leukopenia (Blood and lymphatic system disorders) | 2 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 3 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 3
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 2 | 0
Fatigue (General disorders) | 12 | 2
Pyrexia (General disorders) | 7 | 1
Asthenia (General disorders) | 5 | 0
Oedema peripheral (General disorders) | 3 | 0
Injection site pain (General disorders) | 0 | 1
White blood cell count decreased (Investigations) | 7 | 0
Aspartate aminotransferase increased (Investigations) | 6 | 0
Alanine aminotransferase increased (Investigations) | 4 | 0
Neutrophil count decreased (Investigations) | 4 | 0
Platelet count decreased (Investigations) | 3 | 0
Blood bilirubin increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 8 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Somnolence (Nervous system disorders) | 4 | 0
Lethargy (Nervous system disorders) | 0 | 3
Headache (Nervous system disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0
Insomnia (Psychiatric disorders) | 4 | 0
Vision blurred (Eye disorders) | 2 | 0
Cataract (Eye disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1
Contrast media allergy (Immune system disorders) | 2 | 0
Skin wound (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.